CLINICAL TRIAL: NCT03081273
Title: Corynebacterium Spp Bone and Joint Infection: Retrospective Study of Microbiological, Diagnostic and Therapeutic Features
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0390
Record Dates: First submitted 2017-03-09; First posted 2017-03-16 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Corynebacterium Infections
Keywords: Antimicrobial susceptibility; Biofilm formation; Bone and joint infection; Corynebacterium spp; Osteoblast; Outcome; Prosthetic joint infection
MeSH Terms: conditions — Corynebacterium Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Corynebacterium spp have been considered as innocuous commensals of human skin, but are now accepted as important opportunistic pathogens responsible for various nosocomial infections, especially implicating foreign materials. In particular, they accounted for up to 10% of prosthetic joint infection (PJI), and are mostly identified in chronic forms of bone and joint infections (BJI). However, little is known about the pathophysiological pathway implicated in Corynebacterium BJI, species distribution and antimicrobial susceptibility, and the management of these difficult-to-treat clinical entities.

This study aims to report a retrospective cohort of patients with Corynebacterium spp BJI, aiming to : i) describe microbiological characteristics of the implicated clinical isolates, including species identification and antimicrobial susceptibility (and especially according to previous antimicrobial exposure); ii) assess pathophysiological mechanisms associated with BJI chronicity, including biofilm formation and bone cell invasion, to better understand mechanisms of Corynebacterium spp and to evaluate their ability to distinguished colonizing and infective isolates; iii) describe the medical (nature and duration of antimicrobial therapy) and surgical management of these patients; and iv) evaluate the patient outcome according to this management strategy, and highlight risk factor for treatment failure in order to improve patient's management.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (i.e age ≥ 18-year-old) with microbiologically proven Corynebacterium bone and joint infection, with or without implant

Exclusion Criteria:

* diabetic foot osteomyelitis
* pressure ulcer-associated osteomyelitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with microbiologically proven Corynebacterium bone and joint infection.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Description of microbiological features of Corynebacterium infection | at diagnosis
  microbiological identification at species level will be confirmed for each isolate using routine mass spectrometry (MALDI-TOFF-MS)
antimicrobial susceptibility | at diagnosis
  antimicrobial susceptibility testing performed according to current guidelines of the French committee for antimicrobial susceptibility testing. Antimicrobial susceptibility profile will be interpreted according to previous exposition to antimicrobials, including new molecules such as daptomycin

SECONDARY OUTCOMES:
ability of clinical isolate to form biofilm | at diagnosis
  The ability of clinical isolate to form biofilm will be assessed using the classic photometric method based on crystal violet staining, and the BiofilmRingTest dynamic method evaluating the kinetic of biofilm formation based on magnetic beads immobilization when embedded in biofilm
Corynebacterium isolate ability to invade and persist within bone cells | at diagnosis
  Corynebacterium isolate ability to invade and persist within bone cells will be adressed using an in vitro model of human osteoblastic cells infection, developed in our laboratory, as previously described
Surgical management and antimicrobial therapy in patients with bone or joint infection | at the end of follow up
  Surgical management and antimicrobial therapy will be described and compared to current guidelines
Treatment failure in patients with bone or joint infection | one to two years after the end of antimicrobial therapy
  Treatment failure will include i) clinical and/or microbiological relapse after treatment disruption; ii) the need of additional surgery for septic reason; and iii) death related to the BJI or its management.

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Ferry, MD,PhD, Principal Investigator — Centre de reference des infections ostéo-articulaires de Lyon
Locations (1):
- Centre de reference des infections ostéo-articulaires- Hôpital de la Croix Rousse, Lyon, France

REFERENCES:
- See also: Related Info — http://www.crioac-lyon.fr